CLINICAL TRIAL: NCT03856047
Title: Investigation of Safety and Efficacy of NNC0174-0833 for Weight Management - a Dose Finding Trial.
Brief Title: Research Study Investigating How Well NNC0174-0833 Works in People Suffering From Overweight or Obesity.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4433; U1111-1214-0429 (Other: World Health Organization (WHO)); 2018-001945-14 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: This is a twelve-armed trial comprising of five (0.3, 0.6, 1.2, 2.4 and 4.5 mg OW) of NNC0174-0833 arms and liraglutide 3.0 mg OD arm as active treatment arms and the corresponding 6 placebo arms as comparators. Participants will be randomised 6:1 between the active treatment arms and the placebo arms. The five different NNC0174-0833 placebo arms and the one liraglutide placebo arm will be pooled into one placebo group for statistical analyses of the results.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- NNC0174-0833, 4.5 mg (Experimental): Patients will receive 4.5 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: NNC0174-0833
- NNC0174-0833, 2.4 mg (Experimental): Patients will receive 2.4 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: NNC0174-0833
- NNC0174-0833, 1.2 mg (Experimental): Patients will receive 1.2 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: NNC0174-0833
- NNC0174-0833, 0.6 mg (Experimental): Patients will receive 0.6 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: NNC0174-0833
- NNC0174-0833 0.3 mg (Experimental): Patients will receive 0.3 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: NNC0174-0833
- Placebo 2.4 mg (NNC0174-0833) (Placebo Comparator): Patients will receive 2.4 mg of placebo (NNC0174-0833) once a week as injections for 26 weeks.
  Interventions: Drug: Placebo (NNC0174-0833)
- Placebo 4.5 mg (NNC0174-0833) (Placebo Comparator): Patients will receive 4.5 mg of placebo (NNC0174-0833) once a week as injections for 26 weeks.
  Interventions: Drug: Placebo (NNC0174-0833)
- Placebo 1.2 mg (NNC0174-0833) (Placebo Comparator): Patients will receive 1.2 mg of placebo (NNC0174-0833) once a week as injections for 26 weeks.
  Interventions: Drug: Placebo (NNC0174-0833)
- Placebo 0.6 mg (NNC0174-0833) (Placebo Comparator): Patients will receive 0.6 mg of placebo (NNC0174-0833) once a week as injections for 26 weeks.
  Interventions: Drug: Placebo (NNC0174-0833)
- Placebo 0.3 mg (NNC0174-0833) (Placebo Comparator): Patients will receive 0.3 mg of NNC0174-0833 once a week as injections for 26 weeks.
  Interventions: Drug: Placebo (NNC0174-0833)
- Liraglutide 3.0 mg (Active Comparator): Patients will receive 3.0 mg of liraglutide once daily as injections for 26 weeks.
  Interventions: Drug: Liraglutide 3.0 mg
- Placebo 3.0 mg (Liraglutide) (Placebo Comparator): Patients will receive placebo 3.0 mg(liraglutide) once daily as injections for 26 weeks.
  Interventions: Drug: Placebo (Liraglutide 3.0 mg)

INTERVENTIONS:
Drug: NNC0174-0833 — Participants will get one dose of NNC0174-0833 once weekly. The medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm using NovoPen® 4. Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 26 weeks.
  Arms: NNC0174-0833 0.3 mg; NNC0174-0833, 0.6 mg; NNC0174-0833, 1.2 mg; NNC0174-0833, 2.4 mg; NNC0174-0833, 4.5 mg
Drug: Placebo (NNC0174-0833) — Participants will get one dose of Placebo (NNC0174-0833) once weekly. The medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm using NovoPen® 4. Participants will gradually increase the dose until they reach the target dose, and will continue on the this dose once weekly up to 26 weeks.
  Arms: Placebo 0.3 mg (NNC0174-0833); Placebo 0.6 mg (NNC0174-0833); Placebo 1.2 mg (NNC0174-0833); Placebo 2.4 mg (NNC0174-0833); Placebo 4.5 mg (NNC0174-0833)
Drug: Liraglutide 3.0 mg — Participants will get one dose of liraglutide 3.0 mg once daily. The medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm using pre-filled PDS290 pen-injector. Participants will gradually increase their dose every week until they reach the target dose of 3.0 mg daily. The participants will continue on 3.0 mg of liraglutide, once daily up to 26 weeks.
  Arms: Liraglutide 3.0 mg
Drug: Placebo (Liraglutide 3.0 mg) — Participants will get one dose of Placebo (liraglutide 3.0 mg) once daily. The medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm using pre-filled PDS290 pen-injector. Participants will gradually increase their dose every week until they reach the target dose of 3.0 mg. The participants will continue on Placebo (liraglutide 3.0 mg), once daily up to 26 weeks.
  Arms: Placebo 3.0 mg (Liraglutide)

SUMMARY:
This study will look at the change in body weight in people taking NNC0174-0833, liraglutide and "dummy" medicine, from the start to the end of the study. As well as taking the medicine, participants will have talks with study staff about healthy food choices, how to be more physically active and what participants can do to lose weight. Participants will either take NNC0174-0833, liraglutide or "dummy" medicine - which treatment participants get is decided by chance. Participants will need to take one injection once a week or once a day, depending on the treatment. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. The study will last for about 8 months. Participants will have 12 clinic visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of signing the informed consent.
* Female subject of non-childbearing potential or Male subject who is surgically sterilised (vasectomy) or who is willing to use adequate contraceptive methods (as required by local regulation or practice) throughout the trial (until 'end of trial').
* BMI equal to 30.0 kg/m^2 or greater or BMI equal to 27.0 kg/m^2 or greater with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension or dyslipidaemia (to be assessed at the investigator's discretion).

Exclusion Criteria:

* HbA1c equal to 48 mmol/mol (6.5 percentage) or greater as measured by the central laboratory at screening.
* A self-reported change in body weight greater than 5 kg (11 lbs) within 90 days prior to screening irrespective of medical records.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (54):
- United States (22):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Encompass Clinical Research, Spring Valley, California
  - Nature Coast Clinical Research, Crystal River, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - South Broward Research LLC, Pembroke Pines, Florida
  - St Johns Center For Clinical Research, Ponte Vedra, Florida
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Centennial Medical Group, Elkridge, Maryland
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Rochester Clinical Research, Inc., Rochester, New York
  - PharmQuest, Greensboro, North Carolina
  - Prestige Clinical Research, Franklin, Ohio
  - Albert J Weisbrot, Mason, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Spectrum Medical Research, LLC, Gaffney, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Holston Medical Group Pc, Bristol, Tennessee
  - Texas Diabetes & Endocinology, Round Rock, Texas
  - Washington Center For Weight Management And Research,Inc., Arlington, Virginia
  - National Clinical Research Inc., Richmond, Virginia
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - C-endo Diabetes & Endocrinology Clinic, Calgary, Alberta
  - C-endo Diabetes & Endocrinology Clinic, Edmonton, Alberta
  - The Wharton Medical Clinic Clinical Trials, Hamilton, Ontario
  - Hamilton Medical Research Group, Hamilton, Ontario
- Denmark (2):
  - Aarhus Universitetshospital Diabetes og Hormonsygdomme, Aarhus N
  - Hvidovre Hospital Endokrinologisk forsknings afsnit 159, Hvidovre
- Finland (4):
  - StudyCor, Jyväskylä
  - Itä-Suomen yliopisto, Kuopio
  - Turku University Hospital, Turku
  - Obesity Research Unit, University of Helsinki
- Clinical Research Centre, St. Vincent's University Hospital,, Dublin, Ireland
- Japan (3):
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Tokyo Center Clinic, Tokyo
  - ToCROM Clinic, Tokyo
- Poland (3):
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych, Bialystok
  - Centrum Medyczne Salvia, Katowice
  - Centrum Zdrowia Metabolicznego, Poznan
- Serbia (2):
  - Endocrinology, Diabetes and Metabolism Diseases Clinic, Belgrade
  - Clin. Centre Vojvodina, Clin. endocr., diab. and met. dis., Novi Sad
- South Africa (5):
  - FARMOVS (Pty) LTD, Bloemfontein, Free State
  - Dr Wilhase's rooms, Boksburg, Gauteng
  - Dr R Dulabh, Johannesburg, Gauteng
  - Dr Vawda's site, Durban, KwaZulu-Natal
  - Dr J Reddy, Durban, KwaZulu-Natal
- United Kingdom (7):
  - The Health Centre, Bradford-on-Avon
  - Southmead Hospital, Bristol
  - WISDEM Centre, Coventry
  - University Hospital Aintree, Liverpool
  - Guys Hospital, London
  - UCL - Obesity, London
  - Clifton Medical Centre, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Lau DCW, Erichsen L, Francisco AM, Satylganova A, le Roux CW, McGowan B, Pedersen SD, Pietilainen KH, Rubino D, Batterham RL. Once-weekly cagrilintide for weight management in people with overweight and obesity: a multicentre, randomised, double-blind, placebo-controlled and active-controlled, dose-finding phase 2 trial. Lancet. 2021 Dec 11;398(10317):2160-2172. doi: 10.1016/S0140-6736(21)01751-7. Epub 2021 Nov 16. PMID 34798060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 57 sites in 10 countries as follows: Canada (5), Denmark (2), Finland (4), Ireland (1), Japan (3), Poland (3), Serbia (5), South Africa (5), United Kingdom (7), United States of America (22).
Pre-assignment Details: Participants were randomized in a 6:1 ratio between the active treatment (cagrilintide and liraglutide) arms and the placebo arms. The five different cagrilintide placebo arms and the one liraglutide placebo arm were pooled into one placebo group in the main analyses. Participants received the treatments as an adjunct to reduced-calorie diet and increased physical activity.
Groups:
- Cagrilintide 0.3 mg: Participants were to receive once weekly subcutaneous (s.c.) injection of 0.3 milligrams (mg) cagrilintide for 26 weeks, using NovoPen® 4 pen-injector.
- Cagrilintide 0.6 mg: Participants were to receive once weekly s.c. injection of 0.6 mg cagrilintide for 26 weeks, using NovoPen® 4 pen-injector.
- Cagrilintide 1.2 mg: Participants were to receive once weekly s.c. injection of cagrilintide for 26 weeks, using NovoPen® 4 pen-injector. Participants initially received 0.6 mg of cagrilintide and the dose was then escalated every other week until the target dose of 1.2 mg was reached: 0.6 mg (week 0) and 1.2 mg (week 2 to week 26).
- Cagrilintide 2.4 mg: Participants were to receive once weekly s.c. injection of cagrilintide for 26 weeks, using NovoPen® 4 pen-injector. Participants initially received 0.6 mg of cagrilintide and the dose was then escalated every other week until the target dose of 2.4 mg was reached: 0.6 mg (week 0), 1.2 mg (week 2), 2.4 mg (week 4 to week 26).
- Cagrilintide 4.5 mg: Participants were to receive once weekly s.c. injection of cagrilintide for 26 weeks, using NovoPen® 4 pen-injector. Participants initially received 0.6 mg of cagrilintide and the dose was then escalated every other week until the target dose of 4.5 mg was reached: 0.6 mg (week 0), 1.2 mg (week 2), 2.4 mg (week 4), 4.5 mg (week 6 to week 26).
- Liraglutide 3.0 mg: Participants were to receive once daily s.c. injection of liraglutide for 26 weeks, using PDS290 pen-injector. Participants initially received 0.6 mg of liraglutide and the dose was then escalated every other week until the target dose of 3.0 mg was reached: 0.6 mg (week 0), 1.2 mg (week 1), 1.8 mg (week 2), 2.4 mg (week 3), 3.0 mg (week 4 to week 26).
- Pooled Placebo: Participants were to receive once weekly / once daily s.c. injection of placebo matched to cagrilintide / liraglutide (0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg or 4.5 mg / 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, 3.0 mg ) for 26 weeks respectively.
Period: Overall Study
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Started | 101 | 100 | 102 | 102 | 101 | 99 | 101
Full Analysis Set | 101 | 100 | 102 | 102 | 101 | 99 | 101
Safety Analysis Set | 101 | 100 | 102 | 102 | 101 | 99 | 101
Completed | 97 | 97 | 98 | 101 | 94 | 95 | 95
Not Completed | 4 | 3 | 4 | 1 | 7 | 4 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 3 | 0 | 2
Not completed — Lost to Follow-up | 4 | 2 | 3 | 1 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomised participants according to the intention-to-treat principle.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo | Total
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 101 | 99 | 101 | 706
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (10.3) | 53.2 (11.0) | 52.1 (8.7) | 52.7 (9.8) | 51.5 (12.7) | 51.5 (9.3) | 51.4 (11.9) | 52.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 62 | 63 | 75 | 56 | 65 | 59 | 436
  Male | 45 | 38 | 39 | 27 | 45 | 34 | 42 | 270
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 4 | 2 | 3 | 5 | 4 | 21
  Not Hispanic or Latino | 99 | 99 | 98 | 100 | 98 | 94 | 97 | 685
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 77 | 75 | 75 | 80 | 83 | 82 | 71 | 543
  Asian | 13 | 14 | 15 | 11 | 9 | 13 | 17 | 92
  Black or African American | 9 | 5 | 8 | 9 | 5 | 0 | 9 | 45
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 1 | 5 | 4 | 2 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight (%)
Description: Change in body weight (%) from week 0 to week 26 is presented. For descriptive analysis and statistical analysis the endpoint was evaluated based on the data from in-trial period and treatment adherent period, respectively. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period. Treatment-adherent: a participant is treatment adherent until the first time of non-adherence defined as: participant has not been dosed with trial product within the prior 14 days; participant has received other weight management drug or bariatric surgery; participant has not reached target dose at a pre-specified week; After the pre-specified evaluation week for the target dose, the participant has not received the target dose ±10% within the prior 14 days.
Time Frame: From baseline (week 0) to week 26
Population: The full analysis set included all randomised participants. Overall number of participants analysed = Number of participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage point of body weight
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 96 | 97 | 98 | 99 | 97 | 95 | 95
Percentage point of body weight | -6.1 (3.9) | -6.9 (5.4) | -8.5 (5.4) | -9.5 (6.2) | -10.8 (5.5) | -8.5 (5.6) | -3.0 (5.2)
Statistical Analysis 1: Comparison: Cagrilintide 0.3 mg vs Pooled Placebo; Week 26 responses were analysed using an analysis of covariance (ANCOVA) model with randomised treatment as factor and baseline (week 0) body weight as covariate. For each treatment arm, multiple (x1000) imputation of intermittend missing data was done using Markov Chain Monte Carlo, followed by sequential regression for monotone missing values of body weight including sex and region as factors; Test type: Superiority; p = 0.0002, ANCOVA; Treatment difference (%-points) = -2.99, 95% CI 2-sided [-4.58 to -1.40], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Cagrilintide 0.6 mg vs Pooled Placebo; Week 26 responses were analysed using an analysis of covariance model with randomised treatment as factor and baseline (week 0) body weight as covariate. For each treatment arm, multiple (x1000) imputation of intermittend missing data was done using Markov Chain Monte Carlo, followed by sequential regression for monotone missing values of body weight including sex and region as factors; Test type: Superiority; p < .0001, ANCOVA; Treatment difference (%-points) = -3.78, 95% CI 2-sided [-5.38 to -2.17], Standard Error of Mean 0.82
Statistical Analysis 3: Comparison: Cagrilintide 1.2 mg vs Pooled Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference (%-points) = -6.07, 95% CI 2-sided [-7.77 to -4.36], Standard Error of Mean 0.87
Statistical Analysis 4: Comparison: Cagrilintide 2.4 mg vs Pooled Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference (%-points) = -6.68, 95% CI 2-sided [-8.28 to -5.09], Standard Error of Mean 0.81
Statistical Analysis 5: Comparison: Cagrilintide 4.5 mg vs Pooled Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference (%-points) = -7.79, 95% CI 2-sided [-9.42 to -6.16], Standard Error of Mean 0.83
Statistical Analysis 6: Comparison: Liraglutide 3.0 mg vs Pooled Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < .0001, ANCOVA; Treatment difference (%-points) = -5.98, 95% CI 2-sided [-7.61 to -4.35], Standard Error of Mean 0.83
Statistical Analysis 7: Comparison: Cagrilintide 0.3 mg vs Liraglutide 3.0 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0003, ANCOVA; Treatment difference (%-points) = 2.99, 95% CI 2-sided [1.38 to 4.60], Standard Error of Mean 0.82
Statistical Analysis 8: Comparison: Cagrilintide 0.6 mg vs Liraglutide 3.0 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0082, ANCOVA; Treatment difference (%-points) = 2.20, 95% CI 2-sided [0.57 to 3.84], Standard Error of Mean 0.83
Statistical Analysis 9: Comparison: Cagrilintide 1.2 mg vs Liraglutide 3.0 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.9209, ANCOVA; Treatment difference (%-points) = -0.09, 95% CI 2-sided [-1.82 to 1.64], Standard Error of Mean 0.88
Statistical Analysis 10: Comparison: Cagrilintide 2.4 mg vs Liraglutide 3.0 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3960, ANCOVA; Treatment difference (%-points) = -0.70, 95% CI 2-sided [-2.33 to 0.92], Standard Error of Mean 0.83
Statistical Analysis 11: Comparison: Cagrilintide 4.5 mg vs Liraglutide 3.0 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0316, ANCOVA; Treatment difference (%-points) = -1.81, 95% CI 2-sided [-3.46 to -0.16], Standard Error of Mean 0.84

2. Secondary Outcome: Percentage of Participants With Weight Loss of ≥ 5% of Baseline Body Weight at 26 Weeks
Description: Percentage of participants who achieved a weight loss of greater than or equal to (≥) 5% of baseline (week 0) body weight at 26 weeks is presented. The numbers presented are predictions from a logistic regression model.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 83 | 82 | 72 | 80 | 80 | 78 | 79
Percentage of participants | 57.47 | 61.98 | 75.84 | 74.12 | 88.74 | 76.16 | 30.90

3. Secondary Outcome: Percentage of Participants With Weight Loss of ≥ 10% of Baseline Body Weight at 26 Weeks
Description: Percentage of participants who achieved a weight loss ≥ 10% of baseline (week 0) body weight at 26 weeks is presented. The numbers presented are predictions from a logistic regression model.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 83 | 82 | 72 | 80 | 80 | 78 | 79
Percentage of participants | 15.28 | 24.06 | 35.79 | 43.97 | 53.49 | 39.43 | 10.44

4. Secondary Outcome: Change in Body Weight (Kg)
Description: Change in body weight (Kg) from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 96 | 97 | 98 | 99 | 97 | 95 | 95
Kilograms (kg) | -6.6 (4.3) | -7.1 (5.6) | -9.0 (6.3) | -10.1 (6.7) | -11.8 (6.8) | -9.1 (6.4) | -3.2 (5.8)

5. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 96 | 97 | 98 | 99 | 97 | 95 | 94
centimeters (cm) | -6.2 (5.0) | -6.2 (5.9) | -7.7 (7.1) | -8.1 (7.1) | -9.5 (6.1) | -7.4 (5.8) | -3.4 (5.7)

6. Secondary Outcome: Change in Total Cholesterol
Description: Change in total cholesterol from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 95 | 99 | 97 | 95 | 94
Milligrams per deciliter (mg/dL) | 3.9 (27.8) | -1.8 (22.1) | -3.1 (24.9) | -2.9 (26.7) | -5.4 (22.1) | -9.4 (26.4) | 0.1 (22.8)

7. Secondary Outcome: Change in High Density Lipoprotein (HDL) Cholesterol
Description: Change in HDL cholesterol from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 95 | 99 | 97 | 95 | 94
mg/dL | 1.5 (6.1) | 1.9 (6.9) | 1.1 (7.3) | 1.8 (5.6) | 2.6 (6.9) | 0.8 (6.3) | 0.1 (7.0)

8. Secondary Outcome: Change in Low Density Lipoprotein (LDL) Cholesterol
Description: Change in LDL cholesterol from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 95 | 99 | 97 | 95 | 94
mg/dL | 5.2 (24.0) | -0.3 (19.6) | -0.5 (19.8) | -0.9 (22.1) | -2.7 (19.2) | -5.4 (22.9) | -1.0 (21.5)

9. Secondary Outcome: Change in Very Low Density Lipoprotein (VLDL) Cholesterol
Description: Change in VLDL cholesterol from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 95 | 99 | 97 | 95 | 94
mg/dL | -2.8 (9.1) | -3.4 (11.9) | -3.6 (14.1) | -3.8 (9.4) | -5.4 (10.2) | -4.9 (8.6) | 0.9 (15.6)

10. Secondary Outcome: Change in Triglycerides
Description: Change in triglycerides from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 95 | 99 | 97 | 95 | 94
mg/dL | -13.29 (47.51) | -16.25 (67.59) | -17.98 (71.24) | -19.24 (47.30) | -30.35 (58.35) | -25.42 (45.40) | 8.17 (103.36)

11. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) (%-Point)
Description: Change in HbA1c (measured as percentage point of HbA1c) from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 93 | 97 | 95 | 99 | 95 | 95 | 94
Percentage point of HbA1c | 0.0 (0.2) | -0.1 (0.2) | -0.1 (0.3) | -0.1 (0.3) | -0.1 (0.2) | -0.3 (0.2) | -0.1 (0.2)

12. Secondary Outcome: Change in HbA1c (mmol/Mol)
Description: Change in HbA1c (measured as millimoles per mole (mmol/mol)) from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 93 | 97 | 95 | 99 | 95 | 95 | 94
mmol/mol | -0.5 (2.4) | -0.6 (2.2) | -0.8 (3.0) | -1.0 (2.9) | -1.2 (2.4) | -2.9 (2.7) | -0.6 (2.7)

13. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) (mmol/L)
Description: Change in FPG (measured as mmol/L)) from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 95 | 94 | 99 | 96 | 94 | 94
mmol/L | 0.0 (0.6) | 0.0 (0.5) | -0.2 (0.5) | 0.0 (0.7) | -0.2 (1.0) | -0.5 (0.7) | 0.0 (0.6)

14. Secondary Outcome: Change in FPG (mg/dL)
Description: Change in FPG (measured as milligrams per decilitre (mg/dL)) from week 0 to week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 95 | 94 | 99 | 96 | 94 | 94
mg/dL | -0.7 (10.1) | -0.6 (8.9) | -3.2 (9.7) | 0.0 (12.0) | -3.7 (18.4) | -9.5 (12.4) | -0.5 (11.7)

15. Secondary Outcome: Change in Fasting Insulin
Description: In the below table, fasting insulin data at week 0 and at week 26 is presented. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: The full analysis set included all randomised participants. Number analysed = Number of participants who contributed to the analysis.
Measure: Mean (Standard Error); unit: Picomoles per liter (pmol/L)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 99 | 99 | 101
Picomoles per liter (pmol/L)
  Week 0 | 103.88 (6.62) | 97.43 (6.73) | 96.44 (5.91) | 90.05 (4.70) | 109.99 (8.23) | 95.80 (5.73) | 105.77 (7.06)
  Week 26: number analyzed (Participants) | 94 | 92 | 92 | 94 | 94 | 88 | 85
  Week 26 | 93.07 (6.44) | 82.98 (5.02) | 79.39 (4.53) | 71.22 (4.04) | 78.67 (5.42) | 79.00 (5.46) | 86.55 (5.59)

16. Secondary Outcome: Percentage Change in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Percentage change in HOMA-IR from week 0 to week 26 is presented. Insulin resistance is a condition in which cells fail to respond to normal actions of hormone in body. HOMA-IR is calculated using a subject's fasting plasma insulin and glucose levels. HOMA-IR = fasting serum insulin (micro international units per milliliter (μU/ml)) × fasting plasma glucose (millimoles per liter (mmol/l)) / 22.5. HOMA-IR scores are classified as follows: less than 1.0: considered Insulin sensitive, 0.5-1.4: considered Healthy, Above 1.8: considered Early insulin resistance; Above 2.7 is considered significant insulin resistance. HOMA-IR score ranges from 0-infinity (no upper limit). Higher the score, higher the level of insulin resistance. Endpoint was evaluated based on data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change of HOMA-IR
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 96 | 94 | 99 | 96 | 93 | 94
Percentage change of HOMA-IR | -0.05 (5.83) | -0.60 (8.42) | -1.09 (3.37) | -0.72 (1.94) | -2.12 (7.32) | -0.91 (2.38) | -0.71 (7.10)

17. Secondary Outcome: Change in Homeostatic Model Assessment of Beta-cell Function (HOMA-beta)
Description: Change between the value of HOMA-beta cell function collected at Week 26 and HOMA-beta cell function collected at Week 0 is presented. The homeostatic model assessment estimates steady state beta cell function as a percentage of a normal reference population (%B). HOMA %B = 20 * insulin (micro international units per milliliter (µIU/mL)) / fasting plasma glucose (millimoles per liter (mmol/L)) - 3.5. HOMA-beta score ranges from minus infinity to infinity (no limits). The higher the score the better beta-cell function for HOMA-beta. The endpoint was evaluated based on the data from in-trial period. In-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of Beta Cell Function
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 95 | 95 | 94 | 96 | 95 | 89 | 93
Percentage of Beta Cell Function | -10.7 (94.1) | -20.0 (136.9) | -18.3 (89.8) | -29.9 (54.8) | -39.7 (101.2) | 16.3 (75.1) | -26.0 (122.6)

18. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant administered or used a medicinal product, whether or not considered related to the medicinal product or usage. All AEs reported here are TEAEs. TEAE is defined as an event that had onset date during the on-treatment period. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From week 0 to week 32
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 101 | 99 | 101
Events | 335 | 291 | 361 | 449 | 460 | 470 | 276

19. Secondary Outcome: Number of Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a clinical trial participant administered or used a medicinal product, whether or not considered related to the medicinal product or usage. Serious AE is an AE that resulted in death, life threatening, persistent or significant incapacity or substantial disruption of ability to conduct normal life functions, hospitalization or prolongation of existing hospitalization, congenital anomaly or birth defect, important medical events that may not result in death, be life threatening, or require hospitalization. All SAEs reported in the below table are TESAEs. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From week 0 to week 32
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Number; unit: Events
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 101 | 99 | 101
Events | 8 | 3 | 8 | 6 | 4 | 4 | 4

20. Secondary Outcome: Number of Participants With Occurrence of Anti-drug Antibodies Towards Cagrilintide
Description: Number of participants with occurrence of anti-drug antibodies towards cagrilintide from randomisation from week 0 to week 32 is presented. The endpoint was evaluated based on the data from in-trial period. The in-trial period was defined as the uninterrupted time interval from date of randomisation to date of last contact with trial site. Follow-up time for positive antibodies was not included in the in-trial period. This endpoint is applicable only for the cagrilintide treatment arms.
Time Frame: From week 0 to week 32
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 101
Participants | 51 | 54 | 52 | 75 | 75

21. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured in a sitting position after 5 minutes of rest. The end point is evaluated while the subject is treatment-adherent. A participant is treatment adherent until the first time of non-adherence defined as: a) the participant has not been dosed with trial product within the prior 14 days; b) the participant has received other weight management drug or bariatric surgery c) the participant has not reached target dose at a pre-specified week d) After the pre-specified evaluation week for the target dose, the participant has not received the target dose +/- 10 % within the prior 14 days. This endpoint is applicable only for the cagrilintide treatment arms.
Time Frame: From baseline (week 0) to week 26
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment. Overall number of participants analysed = Number of participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Pooled Placebo
Number analyzed (Participants) | 63 | 63 | 58 | 66 | 68 | 47
millimeter of mercury (mmHg) | -2.2 (5.9) | 0.8 (5.0) | -1.3 (6.0) | -1.2 (5.5) | -1.8 (6.3) | -2.6 (5.5)

22. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: as for outcome 21
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Pooled Placebo
Number analyzed (Participants) | 63 | 63 | 58 | 66 | 68 | 47
mmHg | -4.9 (8.7) | -0.9 (8.1) | -4.9 (9.7) | -5.0 (8.4) | -6.2 (8.5) | -3.8 (7.1)

23. Secondary Outcome: Change in Pulse
Description: Change in pulse from week 0 to week 26 is presented. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 94 | 91 | 92 | 94 | 95 | 88 | 86
beats per minute | -2.1 (8.4) | -0.6 (8.4) | -1.2 (9.1) | -2.0 (10.2) | -4.5 (9.2) | 1.6 (9.1) | -0.1 (8.5)

24. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)
Description: In the below table, hsCRP data at week 0 and at week 26 is presented. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From baseline (week 0) to week 26
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment. Number analysed = Number of participants who contributed to the analysis.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 101 | 99 | 101
milligrams per liter (mg/L)
  Week 0 | 4.5 (6.7) | 4.6 (3.9) | 4.5 (5.8) | 5.8 (7.2) | 5.4 (7.5) | 4.7 (4.1) | 4.6 (6.0)
  Week 26: number analyzed (Participants) | 94 | 92 | 92 | 94 | 94 | 88 | 85
  Week 26 | 3.5 (3.5) | 3.4 (3.0) | 4.6 (8.8) | 4.0 (5.5) | 3.4 (4.0) | 3.5 (3.4) | 3.9 (5.3)

25. Secondary Outcome: Change in Plasminogen Activator Inhibitor-1 (PAI-1) Activity
Description: Due to the assay development issue faced by the laboratory, the Plasminogen Activator Inhibitor-1 (PAI-1) activity (mg/L) was not performed in the study.
Time Frame: From baseline (week 0) to week 26
Population: The safety analysis set included all randomised participants exposed to at least one dose of randomised treatment.
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Change in Renin Activity
Description: Change in renin activity from week 0 to week 26 is presented. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: nanograms per milliliter per hour
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 89 | 92 | 92 | 92 | 91 | 84 | 84
nanograms per milliliter per hour | 2 (12) | 0 (4) | 1 (9) | 1 (10) | 1 (8) | 0 (5) | 0 (5)

27. Secondary Outcome: Change in Aldosterone
Description: Change in aldosterone from week 0 to week 26 is presented. The endpoint was evaluated based on the data from on-treatment period which started from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Time Frame: From baseline (week 0) to week 26
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 94 | 92 | 92 | 94 | 94 | 88 | 85
nanograms per deciliter (ng/dL) | 0.8 (5.4) | 0.8 (6.3) | 0.7 (5.2) | 2.2 (7.1) | 1.1 (5.9) | 1.0 (8.2) | 0.5 (5.1)

ADVERSE EVENTS:
Time Frame: From week 0 to week 32 Results are based on the safety analysis set which included all randomised participants exposed to at least one dose of randomised treatment.
Description: All presented adverse events are treatment emergent adverse events (TEAEs). TEAE is defined as an event that had onset date during the on-treatment period. On-treatment period was from the date of first trial product administration to date of last trial product administration excluding potential off-treatment time intervals triggered by at least 6 consecutive missed doses for cagrilintide or 6 consecutive weeks of missed dosing with liraglutide.
Groups:
- Placebo Pool: Participants were to receive once weekly / once daily s.c. injection of placebo matched to cagrilintide / liraglutide (0.3 mg, 0.6 mg, 1.2 mg, 2.4 mg or 4.5 mg / 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, 3.0 mg ) for 26 weeks respectively.
Arm/Group | Cagrilintide 0.3 mg | Cagrilintide 0.6 mg | Cagrilintide 1.2 mg | Cagrilintide 2.4 mg | Cagrilintide 4.5 mg | Liraglutide 3.0 mg | Placebo Pool
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100 | 0/102 | 0/102 | 0/101 | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 6/101 | 2/100 | 7/102 | 3/102 | 4/101 | 4/99 | 3/101
Other Adverse Events (participants affected / at risk) | 59/101 | 58/100 | 72/102 | 62/102 | 76/101 | 65/99 | 45/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cagrilintide 0.3 mg (N=101) | Cagrilintide 0.6 mg (N=100) | Cagrilintide 1.2 mg (N=102) | Cagrilintide 2.4 mg (N=102) | Cagrilintide 4.5 mg (N=101) | Liraglutide 3.0 mg (N=99) | Placebo Pool (N=101)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cagrilintide 0.3 mg (N=101) | Cagrilintide 0.6 mg (N=100) | Cagrilintide 1.2 mg (N=102) | Cagrilintide 2.4 mg (N=102) | Cagrilintide 4.5 mg (N=101) | Liraglutide 3.0 mg (N=99) | Placebo Pool (N=101)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 6 (7) | 2 (2) | 5 (5) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 5 (5) | 4 (5) | 3 (4) | 5 (5) | 4 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 4 (4) | 2 (2) | 7 (9) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6) | 3 (3) | 6 (7) | 6 (6) | 2 (4) | 7 (8)
Constipation (Gastrointestinal disorders) | 11 (12) | 9 (9) | 8 (8) | 17 (17) | 21 (25) | 26 (30) | 7 (10)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 9 (9) | 8 (8) | 13 (13) | 17 (18) | 9 (10) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 15 (22) | 10 (12) | 8 (9) | 18 (20) | 7 (9) | 18 (28) | 9 (10)
Dizziness (Nervous system disorders) | 8 (10) | 2 (2) | 8 (9) | 9 (14) | 9 (12) | 5 (11) | 3 (7)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 5 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3) | 3 (3) | 4 (4) | 10 (10) | 4 (4)
Fatigue (General disorders) | 8 (8) | 5 (5) | 8 (9) | 10 (12) | 20 (21) | 8 (8) | 3 (3)
Headache (Nervous system disorders) | 10 (15) | 5 (5) | 11 (13) | 11 (17) | 7 (10) | 13 (24) | 12 (22)
Injection site erythema (General disorders) | 5 (5) | 4 (5) | 6 (6) | 7 (23) | 17 (22) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 5 (6) | 2 (2) | 4 (4) | 7 (11) | 7 (7) | 3 (3) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0) | 6 (8) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 4 (26) | 4 (10) | 7 (30) | 12 (44) | 10 (39) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 9 (12) | 13 (14) | 4 (7) | 3 (3) | 10 (12) | 10 (12)
Nausea (Gastrointestinal disorders) | 20 (26) | 27 (32) | 37 (45) | 32 (41) | 47 (61) | 39 (56) | 18 (26)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 3 (4) | 6 (7) | 2 (2) | 6 (7) | 7 (8) | 3 (5)
Urinary tract infection (Infections and infestations) | 1 (1) | 7 (9) | 3 (3) | 4 (5) | 2 (2) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 6 (7) | 5 (5) | 9 (11) | 8 (8) | 20 (31) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03856047/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT03856047/SAP_001.pdf